CLINICAL TRIAL: NCT06165926
Title: Efficacy of Intra-Articular Hypertonic Dextrose Injection and Physical Therapy for Frozen Shoulder: A Randomized Controlled Trial
Brief Title: Hypertonic Dextrose Injection and Physical Therapy for Frozen Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chih-Ya Chang, Doctor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A202305063
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Frozen Shoulder
Keywords: Frozen Shoulder; hypertonic dextrose injection; hydrodilation
MeSH Terms: conditions — Bursitis | interventions — Saline Solution; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15% hypertonic dextrose and physical therapy (Experimental): The patient receives a single ultrasound-guided injection of 15% hypertonic dextrose into the shoulder joint (3 ml of 50% Dextrose + 1 ml of 2% xylocaine + 6 ml of normal saline). Subsequent evaluations occur at the second and fourth weeks, followed by a second round of ultrasound-guided shoulder joint injection treatment, totally two sessions. Simultaneously, the patient undergoes an 8-week physical therapy program, attending sessions twice a week. Each session, lasting approximately 30 minutes, includes joint activities, stretching, and muscle-strengthening exercises under the guidance and supervision of a physical therapist.
  Interventions: Drug: 15% hypertonic dextrose; Other: physical therapy
- normal saline and physical therapy (Placebo Comparator): The patient undergoes a single ultrasound-guided normal saline injection for shoulder joint distension (1 ml of 2% xylocaine + 9 ml of normal saline). Subsequent assessments occur at the second and fourth weeks, followed by a second round of ultrasound-guided shoulder joint injection treatment, totally two sessions. Simultaneously, the patient is undergoing an 8-week physical therapy program, with sessions held twice a week. Each session, lasting approximately 30 minutes, includes joint activities, stretching, and muscle-strengthening exercises under the guidance and supervision of a physical therapist.
  Interventions: Drug: Normal saline; Other: physical therapy

INTERVENTIONS:
Drug: 15% hypertonic dextrose — The solution is prepared with 3 ml of 50% Dextrose, 1 ml of 2% xylocaine, and 6 ml of normal saline.
  The ultrasound-guided injection of 15% hypertonic dextrose is performed at the first week. Subsequent ultrasound-guided shoulder joint injection treatment with hypertonic dextrose is performed at the fourth weeks. A total of 2 sessions of hypertonic dextrose injections are performed.
  Arms: 15% hypertonic dextrose and physical therapy
Drug: Normal saline — The solution is prepared with 1 ml of 2% xylocaine + 9 ml of normal saline. The ultrasound-guided injection of Normal saline(0.9%) is performed at the first week. Subsequent ultrasound-guided shoulder joint injection treatment with Normal saline is performed at the fourth weeks. A total of 2 sessions of Normal saline injections are performed.
  Arms: normal saline and physical therapy
Other: physical therapy — Under the guidance and supervision of a physical therapist, the patient undergoes physical therapy sessions twice a week for a total duration of 8 weeks. Each session lasts approximately 30 minutes and includes joint activities, stretching, and muscle-strengthening exercises.

SUMMARY:
The aim of our study is to investigate whether the combination of hypertonic dextrose injection and shoulder joint hydrodilation, in conjunction with physical therapy, can effectively enhance shoulder joint pain relief, improve range of motion, and enhance daily life functionality in patients with frozen shoulder.

DETAILED DESCRIPTION:
Frozen shoulder (FS), also known as adhesive capsulitis, is a common shoulder ailment, with an annual incidence of approximately 2.4 individuals per 100,000, accounting for about 2% of the total population. The onset of symptoms is predominant in individuals aged forty to sixty years, presenting as persistent restrictions in shoulder joint mobility accompanied by shoulder joint pain.

While the detailed mechanisms underlying frozen shoulder remain unclear, arthroscopic examination of the shoulder joint reveals thickening and contraction of the shoulder joint capsule, adhesion with the humeral head, and a reduction in joint cavity volume, particularly in the folds of the axillary recess of the joint capsule and its surrounding areas. These changes contribute to restricted shoulder joint mobility in individuals with frozen shoulder. Additionally, research suggests that in cases of severe inflammation, certain cytokines and growth factors drive fibroblasts to replace normal tissue through repair and remodeling responses. This excessive fibrosis and the loss of normal collagen remodeling response further contribute to the development of frozen shoulder.

The meta-analysis published in JAMA Network in 2020 highlighted the significance of medium to long-term physical therapy in facilitating subsequent improvements in range of motion and functionality for patients with adhesive capsulitis, also known as frozen shoulder. Moreover, numerous studies suggest that combining intra-articular injections with shoulder joint capsular distension procedures, such as hydrodilatation, can enhance shoulder joint function and mobility.

Prolotherapy is a non-surgical regenerative injection therapy involving the injection of a solution into painful or degenerated areas. The injected proliferants induce a local inflammatory response, triggering the release of growth factors and stimulating fibroblasts and collagen-producing cells. This process mimics the natural healing mechanisms of the body, promoting cellular tissue growth through a beneficial inflammatory response. In clinical practice, the most commonly utilized solution for prolotherapy is the hypertonic dextrose with concentrations ranging from 15% to 25%. Concentrations exceeding 10% are generally considered to induce local inflammation, thereby triggering a cascade of reparative effects.

Although there have been numerous studies on shoulder joint capsular distension procedures in the past, the injected solutions often consisted of corticosteroids and saline. In clinical observations, the use of hypertonic dextrose injection combined with shoulder joint capsular distension appears to offer improved outcomes in terms of pain relief and joint angle progression in patients with adhesive capsulitis. However, there is currently no research investigating the effectiveness of hypertonic dextrose injection combined with shoulder joint capsular distension for treating frozen shoulder. Therefore, this study represents the first exploration of whether the use of hypertonic dextrose injection combined with shoulder joint hydrodilatation and physical therapy is more effective than the conventional approach using saline injection combined with physical therapy in the treatment of frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. Frozen shoulder is diagnosed by physicians based on the patient's medical history, physical examination, X-ray, and ultrasound reports.
2. The symptoms persist for more than 3 months.
3. There is a reduction of at least 30 degrees in at least two of the affected shoulder joint angles compared to the angles of the healthy side: shoulder flexion, abduction, and external rotation.

Exclusion Criteria:

1. Ultrasound of the shoulder muscles reveals a complete tear or massive tear of the rotator cuff tendon or calcific tendinitis.
2. Systemic rheumatic disease.
3. Previous shoulder fracture or surgical intervention.
4. Recent shoulder joint injections within the last 3 months.
5. Acute cervical nerve root compression.
6. Current pregnancy or breastfeeding.
7. Poorly controlled diabetes (intravenous glucose injection may cause temporary blood sugar elevation).
8. Patients with cancer.
9. Cognitive impairment, inability to follow simple instructions, or inability to cooperate with the study procedures.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | the change from baseline, post-intervention 2, 4, 8, 12 weeks and 6 months
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. "0" means painless and "10" means extremely painful.

SECONDARY OUTCOMES:
Range of Motion (ROM) | the change from baseline, post-intervention 2, 4, 8, 12 weeks and 6 months
  Using a standardized goniometer, passive shoulder joint range of motion angles on the affected side are measured in standard positions, including flexion, extension, abduction, external rotation, and internal rotation.
Shoulder Pain and Disability Index (SPADI) | the change from baseline, post-intervention 2, 4, 8, 12 weeks and 6 months
  Shoulder function and disability were evaluated using the Chinese version of the Shoulder Pain and Disability Index (SPADI), a self-report questionnaire that yields pain and disability domain and total scores. The SPADI includes five questions on pain and eight questions on disability, referring to various problems with the shoulder encountered over the preceding week. Each item's score ranges from 0 (no pain/normal) to 10 (maximal pain/disability), with total scores of pain from 0-50 and disability from to 0-80. A higher score shows more disability.